CLINICAL TRIAL: NCT01045642
Title: Open Label Balanced Randomized,Two-treatment,Two-period,Two-sequence,Single Dose,Crossover Oral Bioequivalence Study of Omeprazole Mg 20mg DR Capsules With Prilosec OTCTM 20mg in 38 Healthy,Adult,Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Omeprazole Magnesium 20 mg DR Capsules Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sr. Director - R&D, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OMP/CR/070/0607
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Bioequivalence; Omeprazole; Crossover
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prilosec 20 mg Tablets (Active Comparator)
  Interventions: Drug: Omeprazole
- Omeprazole Magnesium DR 20 mg Capsules (Experimental)
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — Omeprazole Magnesium DR Capsules 20 mg
  Other Names: Prilosec OTC 20 mg Tablets

SUMMARY:
An open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose, crossover oral bioequivalence study of Omeprazole Magnesium 20 mg DR Capsules of Dr. Reddy's Laboratories Limited, India and Prilosec OTCTM 20 mg (Omeprazole Magnesium DR Tablets) of Procter and Gamble, Cincinnati, Sweden in 38 healthy, adult, human subjects under fasting conditions.

DETAILED DESCRIPTION:
All study related procedures, restrictions, duration, dates and timings, information on the study formulation and confidentiality of subject data were explained clearly to the volunteers by clinical personnel at the time of obtaining informed consent. Volunteers who signed the consent form and showed"their willingness to participate in the study were enrolled. Volunteers who satisfied the inclusion and exclusion criteria and found to be healthy on physical examination with laboratory investigation values within reference limits were considered eligible to be admitted into the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who provided written informed consent.
* Subjects who were healthy adults within 18-45 years of age (inclusive).
* Body mass index of ≥ 18 kg/m2 and ≤ 25 kglm2 with body weight not less than 50 kg.
* Subjects who had normal health as determined by medical history and physical examination performed within 15 days prior to the dosing of Period-I.
* Had normal ECG, Chest X-ray and vital signs.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.
* If subject is a female volunteer and is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device(IUD), or abstinence, or is postmenopausal for at least 1 year, or is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)
* Each female subject will be given a urine pregnancy test at check-in for period-I, period-II and post study.

Exclusion Criteria:

* Subjects incapable of understanding the informed consent.
* Subjects with BP≤90/60 mrn/Hg or BP≥140/90 mrn/Hg
* History of hypersensitivity or idiosyncratic reaction to Omeprazole or any other related drug.
* Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function. Subjects with a history of tuberculosis, epilepsy, asthma(during past 5 years),diabetes, psychosis or glaucoma will not be eligible for the study
* Regular smoker who smokes more than ten cigarettes daily and has difficulty in abstaining from smoking for the duration of each study period.
* Subjects who has taken over the counter or prescribed medications, including any enzyme modifying drugs or any systemic medication within the past 30 days prior to dosing in Period-1.
* History of any psychiatric illness, which may impair the ability to provide written, informed consent.
* Subjects who have a history of alcohol or substance abuse within the last 5 years
* Subjects with clinically significant abnormal values of laboratory parameters.
* Subjects who have participated in any other clinical investigation using experimental drug or had bled more than 350 mL in the past 3 months.
* Subjects who have used any drugs or substances known to be strong inhibitors of CYP enzymes (formerly known as cytochrome P450 enzymes) within 28 days prior to the first dose.
* Subjects who have used any drugs or substances known to be strong inducers of CYP enzymes (formerly known as cytochrome P450 enzymes) within 28 days prior to the first dose.
* Subjects who are unable to or likely to be non-compliant with protocol requirements or restrictions.
* Any subject in whom Omeprazole is contraindicated for medical reasons
* Subjects who are intolerant to venipuncture
* Subjects with positive urine screen for drugs of abuse. All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at each study period check-in. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate
* Female volunteers who has used implanted or injected hormonal contraceptives anytime during the 6 months prior to study or used hormonal contraceptives within 14 days before dosing
* Female volunteers demonstrating a positive pregnancy screen.
* All female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or inconclusive results will be withdrawn from the study
* Female volunteers who are currently breast feeding.
* Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr IS Gandhi, Principal Investigator — Vimta Labs Limited
Locations (1):
- Vimta Labs Limited, Hyderabad, Andhra Pradesh, India